CLINICAL TRIAL: NCT04378933
Title: Glasses for Adolescent Delayed Sleep-Wake Phase Disorder (GLAD)
Brief Title: Glasses for Adolescent Delayed Sleep-Wake Phase Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, R. Robert Auger, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-003036
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Delayed Sleep-Wake Phase Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Amber Glasses and Fixed Wake (Experimental): Participants will wear glasses with amber lenses beginning 7 hours before average baseline mid-sleep time until the time of intended sleep onset or until a duration of 7 hours of use is reached. Participants will also be required to wake up at the same time (±30 mins).
  Interventions: Device: Amber Glasses
- Clear glasses and Free Wake (Active Comparator): Participants will wear identically appearing glasses with clear lenses beginning 7 hours before average baseline mid-sleep time until the time of intended sleep onset or until a duration of 7 hours of use is reached. Participants will not be given instructions regarding sleep schedule.
  Interventions: Device: Clear Lens Glasses

INTERVENTIONS:
Device: Amber Glasses — Half of the participants will be wearing the amber glasses to see if they can help with sleep onset.
  Arms: Amber Glasses and Fixed Wake
Device: Clear Lens Glasses — Half of the participants will be wearing the clear glasses to see if the glasses help with sleep onset.
  Arms: Clear glasses and Free Wake

SUMMARY:
The purpose of this study is to determine if evening amber glasses combined with stable wake times will show an increase in total sleep time (TST) and an advance in sleep onset times (shift earlier) compared to the control group.

DETAILED DESCRIPTION:
We propose a 3-week field study that examines the efficacy, acceptance, and compliance of using evening amber glasses to block evening light combined with a stable wake time in adolescents (14-17 years) with DSWPD (International Classification of Sleep Disorders [ICSD-3] criteria).3 After 1 week of baseline measurements, subjects will be instructed to wear glasses (which allow 14% entry of ambient light exposure) starting 7 h before individually calculated midsleep time measured during the preceding week. This corresponds to the time when adolescents are most sensitive to phase delaying light according to Co-I Crowley's recently published phase response curve (PRC) to light in adolescents (Figure 1).22 This "amber glasses + stable wake time" group will be compared to a control group: adolescent DSWPD patients who will wear clear-lensed glasses (which allow 100% of ambient light to reach the eyes, otherwise identical in appearance) in the evening at the same times as the alternate group, but without scheduled wake times. Outcome measures will include TST and sleep onset time derived from wrist actigraphy, daytime subjective sleepiness, salivary DLMO, and assessments of acceptance and compliance.

ELIGIBILITY:
Inclusion Criteria

* Regular school attendance in the setting of a fixed start time.
* Adherence to ICSD-3 DSWPD diagnostic criteria.
* Average spontaneous weekend wake time ≥1 hour than school day wake time.
* Initiation of school-night sleep at 12 a.m. or later, ≥50% of the time, during a 14-day period (items 3-4 to be determined by sleep logs and actigraphy). As there are no discrete clock times associated with the ICSD-3 DSWPD description, this cutoff is based on data obtained from the 2006 Sleep in America Poll and experiences gleaned from prior recruitment.

Exclusion Criteria

* A positive urine drug abuse screen will disqualify the individual from further participation.
* Subjects will be withdrawn from the study if the sleep log and wrist monitor activity does not correspond with the sleep schedule identified with the pre-study sleep log.
* Alcohol and nicotine use will also be screened to qualify for the study. We will also screen for alcohol immediately before each DLMO assessment because alcohol acutely suppresses melatonin.
* Patients receiving medications that might contribute to sleep disturbances and/or affect treatment responses will be considered ineligible (e.g., hypnotics, antidepressants, stimulants, non-steroidal anti-inflammatory drugs (NSAIDs), beta blockers).
* All subjects will be asked to refrain from caffeine use on the days of phase assessments, and to cease ingestion at least 6 hours prior to nightly bedtime.
* The Ishihara Color Blindness Test will be done and patients who are color blind/deficient will be disqualified from participating in the study.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Robert Auger, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Amber Glasses and Fixed Wake: Participants wore glasses with amber lenses beginning 7 hours before average baseline mid-sleep time until the time of intended sleep onset or until a duration of 7 hours of use was reached. Participants were also required to wake up at the same time (±30 mins).
  Amber Glasses: Half of the participants wore the amber glasses to see if the glasses helped with sleep onset.
- Clear Glasses and Free Wake: Participants wore identically appearing glasses with clear lenses beginning 7 hours before average baseline mid-sleep time until the time of intended sleep onset or until a duration of 7 hours of use was reached. Participants were given instructions regarding sleep schedule.
  Clear Lens Glasses: Half of the participants wore clear glasses to see if the glasses helped with sleep onset.
Period: Overall Study
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (1.2) | 16.8 (1.2) | 16.6 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 9 | 13 | 22
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in School Night Sleep Onset Time
Description: The time in hours that sleep onset time shifted earlier during school nights. Measured by self-reporting logs and a wrist actigraphy that detects when subjects are active or sleeping.
Time Frame: baseline, week 3
Population: Data not collected nor analyzed for 10 subjects in Amber arm and 9 subjects in Clear arm
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
Number analyzed (Participants) | 7 | 8
hours | 0.4 (1.3) | 0.6 (1.0)

2. Primary Outcome: Change in Non-school Night Sleep Onset Time
Description: The time in hours that sleep onset time shifted earlier during non-school nights. Measured by self-reporting logs and a wrist actigraphy that detects when subjects are active or sleeping.
Time Frame: baseline, week 3
Population: Data not collected nor analyzed for 10 subjects in Amber arm and 9 subjects in Clear arm
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
Number analyzed (Participants) | 7 | 8
hours | 1.1 (1.0) | 0.03 (1.0)

3. Primary Outcome: Change in Dim Light Melatonin Onset (DLMO)
Description: The time of day the subject feels sleepy during the overnight lab stays. It is a marker of biological time. Data are provided in decimal and military time (e.g., 10:00 pm equals 22.00).
  Using a light lux meter, the lighting in the room was limited to no more than 5 lux of light. Measured by self-reported logs and a wrist actigraphy that detects when subjects are active or sleeping.
Time Frame: baseline, week 3
Population: Data not collected nor analyzed for 10 subjects in Amber arm and 9 subjects in Clear arm
Measure: Mean (Standard Deviation); unit: decimal military time
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
Number analyzed (Participants) | 7 | 8
decimal military time
  baseline | 21.51 (1.55) | 22.36 (2.18)
  week 3 | 21.11 (1.12) | 23.05 (2.17)

4. Primary Outcome: Change in Dim Light Melatonin Onset (DLMO) Phase Shift
Description: The time in hours the circadian clock shifted the sleep onset time. Using a light lux meter, the lighting in the room will be limited to no more than 5 lux of light. Measured by self-reported logs and a wrist actigraphy that detects when subjects are active or sleeping.
Time Frame: baseline, week 2
Population: Data not collected nor analyzed for 10 subjects in Amber arm and 9 subjects in Clear arm
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
Number analyzed (Participants) | 7 | 8
hours | 1.0 (2.0) | 0.4 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each subject from baseline to end of study, approximately 3 weeks
Arm/Group | Amber Glasses and Fixed Wake | Clear Glasses and Free Wake
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT04378933/Prot_SAP_001.pdf